CLINICAL TRIAL: NCT07178197
Title: Association of Sarcopenia With Quality of Life and Progression of Disease in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Sarcopenia in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Sibel Naycı, Prof. Dr., Mersin University
Other Study IDs: 2022/736
Record Dates: First submitted 2025-08-25; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF); Sarcopenia
Keywords: idiopathic pulmonary fibrosis; sarcopenia; skeletal muscle mass index; bioelectrical impedance analysis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- idiopathic pulmonary fibrosis (IPF): The prevalence of sarcopenia was investigated in patients with IPF who met the inclusion and exclusion criteria. The relationship between sarcopenia and quality of life and disease progression in patients with IPF was evaluated.

SUMMARY:
Sarcopenia negatively affects the prognosis of chronic diseases. However, the importance of sarcopenia in patients with idiopathic pulmonary fibrosis (IPF) has been less emphasized. The aim of the study is to determine the prevalence of sarcopenia in patients with IPF and to evaluate the impact of sarcopenia on quality of life and disease progression.

This study was designed as a descriptive cross-sectional. The study included patients diagnosed with IPF. Hand dynamometry and bioelectrical impedance analysis (BIA) were used to for diagnose of sarcopenia. Pulmonary function tests, maximal inspiratory pressure (MIP), and maximal expiratory pressure (MEP) measurements were examined. The 6-minute walk distance (6MWD) and 4-meter walking speed were recorded. The St. George Respiratory Questionnaire (SGRQ) was used to assess quality of life. All patients were evaluated for progressive disease.

DETAILED DESCRIPTION:
The study was designed as a cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Signing the informed consent form
* Having a diagnosis of IPF for at least one month

Exclusion Criteria:

* Pregnancy
* History of cancer within the last 5 years
* History of lung surgery
* History of neuromuscular disease
* Active pulmonary tuberculosis
* Active respiratory tract infection
* Inability to perform pulmonary function tests
* Presence of a pacemaker
* History of systemic steroid use within the past 3 months
* Inability to use a hand dynamometer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the study were those diagnosed with IPF according to the ATS/ERS/JRS/ALAT 2022 guidelines and who applied to the Department of Pulmonary Diseases at Mersin University Faculty of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Hand Grip Strength | through study completion, an average of 1 year
  Hand Grip Strength (kg)- Grip strength measurement using a hand dynamometer
SMI (skeletal muscle mass index) | through study completion, an average of 1 year
  SMI (skeletal muscle mass index) (kg/m2) - SMI measurement using the Bioelectrical Impedance Analysis (BIA) device
Forced Expiratory Volume in 1 second (FEV1) | through study completion, an average of 1 year
  Measurement of FEV1 for the assessment of pulmonary function
Forced Vital Capacity (FVC) | through study completion, an average of 1 year
  Measurement of FVC for the assessment of pulmonary function
Diffusing Capacity of The Lungs for Carbon Monoxide (DLCO) | through study completion, an average of 1 year
  Measurement of DLCO for the assessment of pulmonary function.
Total Lung Capacity (TLC) | through study completion, an average of 1 year
  Measurement of TLC for the assessment of pulmonary function.
Respiratory Muscle Strength | through study completion, an average of 1 year
  Measurement of maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) for assessment of respiratory muscle strength
Six Minute Walk Test (6MWT) | through study completion, an average of 1 year
  Distance walked in six minutes (m)
Gait speed | through study completion, an average of 1 year
  4-meter walking speed (m/s)
St. George's Respiratory Questionnaire (SGRQ) | through study completion, an average of 1 year
  The questionnaire is designed to measure quality of life. It consists of symptom, activity, impact, and total scores. Each score ranges from 0 to 100. High scores indicate lower quality of life.
Progressive Disease | through study completion, an average of 1 year
  Examination of all participants from clinical, physiological, and radiological perspectives

SECONDARY OUTCOMES:
Body Mass Index ( BMI) | through study completion, an average of 1 year
  kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University Faculty of Medicine, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No